CLINICAL TRIAL: NCT00012987
Title: Implementing Guidelines for Smoking Cessation: A Randomized Trial of Evidence-Based Quality Improvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPG 97-002
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Smoking; Smoking Cessation; Quality Improvement
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Quality Improvement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Quality Improvement

INTERVENTIONS:
Behavioral: Quality Improvement

SUMMARY:
Smoking is a serious and common health risk among veterans. Given the press of national initiatives and local incentives to improve smoking cessation care in response to VA performance measures, this study tests a widely applicable approach to clinical practice guidelines implementation, namely evidence-based quality improvement, which is directly relevant to the translation of efficacious treatments into enhancements in VA health care policy and practice. Evidence-Based Quality Improvement (EBQI) focuses on improved provider adherence to smoking cessation guidelines and a decrease in patient smoking rates in a manner designed to produce short- and long-term health improvements and cost benefits at the organizational level.

DETAILED DESCRIPTION:
Background:

Smoking is a serious and common health risk among veterans. Given the press of national initiatives and local incentives to improve smoking cessation care in response to VA performance measures, this study tests a widely applicable approach to clinical practice guidelines implementation, namely evidence-based quality improvement, which is directly relevant to the translation of efficacious treatments into enhancements in VA health care policy and practice. Evidence-Based Quality Improvement (EBQI) focuses on improved provider adherence to smoking cessation guidelines and a decrease in patient smoking rates in a manner designed to produce short- and long-term health improvements and cost benefits at the organizational level.

Objectives:

Adherence to smoking cessation guidelines requires practice changes at the patient, provider, and system levels to achieve optimal quit rates. The objective of this study was to evaluate the effectiveness of evidence-based quality improvement (EBQI)�an expert-designed and locally implemented clinical reorganization of smoking cessation care�on changes in smoking cessation (SC) practice among primary care providers and health outcomes among veteran smokers.

Methods:

An evidence-based quality improvement intervention comprising provision of physician and patient educational materials, local priority setting with leadership and providers, and local adaptation of expert-designed protocols was implemented in experimental VA primary care practices (n=9). VA control sites (n=9), matched on size and academic affiliation, received smoking cessation guideline copies. We randomly sampled, consented, screened and surveyed primary care patients at all 18 sites (n=1,941 smokers) and used computer-assisted telephone interviewing to assess sociodemographics, health status, function, and smoking behavior, attitudes and treatment experience. Post-intervention 12-month follow-up interviews were completed using the same measures (n=1,080). We used multiple imputation using hotdeck techniques and applied both enrollment and attrition weights to the patient-level data. We used weighted logistic regression to evaluate intervention effects, controlling for patient-level predictors of quit attempts and quit status (e.g., level of addiction, readiness to change, age, health).

Status:

The project is completed. Analysis is ongoing for manuscripts.

ELIGIBILITY:
Inclusion Criteria:

VA Medical Center or outpatient clinics with at least 3000 patients.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott E Sherman, MD MPH, Principal Investigator — VA Greater Los Angeles Healthcare System, Sepulveda, CA; Elizabeth M. Yano, PhD MSPH, Principal Investigator — VA Greater Los Angeles Healthcare System, Sepulveda, CA
Locations (2):
- United States (2):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA Greater Los Angeles Healthcare System, Sepulveda, CA, Sepulveda, California

REFERENCES:
- [Result] Sherman SE, Yano EM, York LS, Lanto AB, Chernof BA, Mittman BS. Assessing the structure of smoking cessation care in the Veterans Health Administration. Am J Health Promot. 2006 May-Jun;20(5):313-8. doi: 10.4278/0890-1171-20.5.313. PMID 16706001
- [Result] Sherman SE, Fu SS, Joseph AM, Lanto AB, Yano EM. Gender differences in smoking cessation services received among veterans. Womens Health Issues. 2005 May-Jun;15(3):126-33. doi: 10.1016/j.whi.2005.01.001. PMID 15894198
- [Result] Sherman SE, Joseph AM, Yano EM, Simon BF, Arikian N, Rubenstein LV, Parkerton P, Mittman BS. Assessing the institutional approach to implementing smoking cessation practice guidelines in veterans health administration facilities. Mil Med. 2006 Jan;171(1):80-7. doi: 10.7205/milmed.171.1.80. PMID 16532880
- [Result] Jonk YC, Sherman SE, Fu SS, Hamlett-Berry KW, Geraci MC, Joseph AM. National trends in the provision of smoking cessation aids within the Veterans Health Administration. Am J Manag Care. 2005 Feb;11(2):77-85. PMID 15726855
- [Result] Sherman SE, Yano EM, Lanto AB, Simon BF, Rubenstein LV. Smokers' interest in quitting and services received: using practice information to plan quality improvement and policy for smoking cessation. Am J Med Qual. 2005 Jan-Feb;20(1):33-9. doi: 10.1177/1062860604273776. PMID 15782753
- [Result] Meredith LS, Yano EM, Hickey SC, Sherman SE. Primary care provider attitudes are associated with smoking cessation counseling and referral. Med Care. 2005 Sep;43(9):929-34. doi: 10.1097/01.mlr.0000173566.01877.ac. PMID 16116358
- [Result] Sherman SE, Lanto AB, Nield M, Yano EM. Smoking cessation care received by veterans with chronic obstructive pulmonary disease. J Rehabil Res Dev. 2003 Sep-Oct;40(5 Suppl 2):1-12. doi: 10.1682/jrrd.2003.10.0001. PMID 15074449
- [Result] Mojica WA, Suttorp MJ, Sherman SE, Morton SC, Roth EA, Maglione MA, Rhodes SL, Shekelle PG. Smoking-cessation interventions by type of provider: a meta-analysis. Am J Prev Med. 2004 Jun;26(5):391-401. doi: 10.1016/j.amepre.2004.02.014. PMID 15165655
- [Result] Yano EM, Rubenstein LV, Farmer MM, Chernof BA, Mittman BS, Lanto AB, Simon BF, Lee ML, Sherman SE. Targeting primary care referrals to smoking cessation clinics does not improve quit rates: implementing evidence-based interventions into practice. Health Serv Res. 2008 Oct;43(5 Pt 1):1637-61. doi: 10.1111/j.1475-6773.2008.00865.x. Epub 2008 Jun 3. PMID 18522670
- [Result] Lombardero A, Campbell DG, Harris KJ, Chaney EF, Lanto AB, Rubenstein LV. Prevalence and correlates of smoking status among veterans affairs primary care patients with probable major depressive disorder. Addict Behav. 2014 Mar;39(3):538-45. doi: 10.1016/j.addbeh.2013.10.030. Epub 2013 Nov 4. PMID 24290879